CLINICAL TRIAL: NCT02003079
Title: Evaluating the Impact of Chronic Rhinosinusitis on the Health-Related Quality of Life Among Adults With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Hospital, Canada
Other Study IDs: CFSinus-001
Record Dates: First submitted 2013-07-11; First posted 2013-12-06 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Reoperation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Diagnosed with or without Chronic Rhinosinusitis
  Interventions: Behavioral: Cystic Fibrosis Questionnaire (Revised) for Teens/Adults

INTERVENTIONS:
Behavioral: Cystic Fibrosis Questionnaire (Revised) for Teens/Adults

SUMMARY:
Individuals with Cystic Fibrosis (CF) have a defective protein, which is known as the cystic-fibrosis transmembrane regulator (CFTR). The CFTR transports salt and hydrates mucous. CFTR defects may result in the accumulation of thick mucous in the sinus cavities. As a result, the tiny hair-like structures that sweep mucous out of the sinuses cannot function properly, which can lead to recurrent infection and swelling of the sinus walls. When symptoms are persistent for more than 12 weeks, this is known as chronic rhinosinusitis (CRS). The symptoms that are associated with CRS are nasal discharge, congestion, facial pain or pressure and reduced sense of smell. CRS in non-CF patients affects a large number of individuals in Canada and has been found to be associated with poor quality of life. In the CF population the life expectancy is increasing but chronic disease like CRS is becoming increasingly prevalent. Investigators currently do not know the impact that CRS has on the health-related quality of life in adults with CF and how many suffer from symptoms. The investigators aim to determine the impact of CRS among adults with CF, in order to gain a better understanding of chronic disease among these individuals. The investigators strongly feel this research will improve the referral processes between Respirologists and Otolaryngologists, thereby improving treatment and quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Definitive diagnosis of cystic fibrosis from positive genetic or sweat chloride test
* Currently enrolled at the St. Paul's Cystic Fibrosis Clinic

Exclusion Criteria:

* Individuals unable to understand the purpose, methods and conduct of this study.
* Patients unwilling to provide informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals over the age of 19 years with a definitive diagnosis of Cystic Fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Difference in Cystic Fibrosis-specific HRQoL score among those with and without CRS. | One clinic visit (30 minutes)
  Subjects will complete questionnaires meant to assess the severity of their symptoms as a cumulative experience of the last two weeks leading up to the visit. Subjects will also undergo nasal endoscopy examination during the same visit. All of the study procedures and data collection will be completed in one visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amin R Javer, MD FRCSC FARS, Principal Investigator — St Paul's Sinus Center
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Habib AR, Buxton JA, Singer J, Wilcox PG, Javer AR, Quon BS. Association between Chronic Rhinosinusitis and Health-Related Quality of Life in Adults with Cystic Fibrosis. Ann Am Thorac Soc. 2015 Aug;12(8):1163-9. doi: 10.1513/AnnalsATS.201504-191OC. PMID 26011015